CLINICAL TRIAL: NCT03990779
Title: Echocardiography Findings and Perioperative Outcomes in Children Undergoing Congenital Heart Surgery: Prospective Observational Study
Brief Title: Echocardiography Findings and Perioperative Outcomes in Children
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Other Study IDs: H1906-031-1038
Record Dates: First submitted 2019-06-14; First posted 2019-06-19 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Congenital Cardiac Defect
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with congenital cardiac disease: Children with congenital cardiac disease who undergoing surgery
  Interventions: Diagnostic Test: Echocardiography

INTERVENTIONS:
Diagnostic Test: Echocardiography — Echocardiographic examination before and after cardiopulmonary bypass

SUMMARY:
This study evaluates the association between perioperative echocardiographic Doppler findings and clinical outcomes in pediatric patients undergoing cardiac surgery. In our center, anesthesiologists perform transthoracic or transesophageal echocardiography during perioperative period routinely in children undergoing surgery for congenital cardiac disease. Echocardiographic findings include the doppler patterns of hepatic vein, portal vein, renal artery, renal vein and splenic vein before and after cardiopulmonary bypass. Portal pulsatility index, renal resistive index, and respiratory variations in peak aortic blood flow velocity and diameter of inferior vena cava are measured.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients undergoing cardiac surgery

Exclusion Criteria:

* Applying extracorporeal membrane oxygenator prior to surgery
* Trouble applying echocardiography

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Pediatric patients undergoing cardiac surgery
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Characteristics of Doppler values and its derived parameters of portal vein, hepatic vein, renal artery and vein, and splenic vein measured using echocardiography in children with congenital cardiac disease | after anesthetic induction until the end of surgery
  To find the characteristics and standard values of Doppler findings measured by echocardiography before and after congenital cardiac surgery
Association between Doppler values measured by echocardiography and clinical outcomes after pediatric cardiac surgery | through study completion, an average 1-2 years
  To evaluate whether Doppler values of portal vein, hepatic vein, renal artery and vein, and splenic vein measured using echocardiography can predict major adverse outcomes after pediatric cardiac surgery

SECONDARY OUTCOMES:
Number of patients with major adverse outcomes after pediatric cardiac surgery | through study completion, an average 1-2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee JH, Denault AY, Beaubien-Souligny W, Kang P, Kim J, Kim HW, Ji SH, Jang YE, Kim EH, Kim HS, Kim JT. Higher portal venous pulsatility is associated with worse clinical outcomes following congenital heart surgery: a single-centre prospective cohort study. Can J Anaesth. 2023 Dec;70(12):1957-1969. doi: 10.1007/s12630-023-02605-0. Epub 2023 Nov 2. PMID 37919629